CLINICAL TRIAL: NCT00735826
Title: A Clinical Trial to Validate Molecular Targets of Vorinostat in Patients With Aerodigestive Tract Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Konstantin Dragnev, Staff Physician, Hematology-Oncology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D-0828
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Aerodigestive Tract Cancer; Lung Cancer; Esophageal Cancer; Head and Neck Cancer
Keywords: resectable; stage I-III; NSCLC; vorinostat; esophagus; head and neck; proof of principle
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat 400 mg (Experimental): Vorinostat will be administered orally once daily in an open-labeled unblinded manner to all subjects enrolled in the study. Subjects will received 400 mg once daily on a continuous daily basis for 7 to 10 days prior to surgical resection.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Vorinostat will be administered orally once daily in an open-labeled, unblinded manner to all subjects enrolled in the study. Subjects will receive vorinostat 400 mg once daily on a continuous daily basis for 7 to 10 days prior to surgical resection. Vorinostat should be taken with food within 0 to 30 minutes of a meal if possible. Patients should take the medication at approximately the same time each day on an ongoing basis. Missed doses will not be made up.

SUMMARY:
The primary aim is to study the effects of vorinostat on cyclin E, cyclin D1 and Ki-67 expression in aerodigestive tract tumors (lung, esophagus, and head and neck). Secondary aims are: To evaluate the concentration of vorinostat in tumor tissue and to correlate tumor tissue distribution with the plasma level in these patients; to perform exploratory analyses of the effects of vorinostat on the induction of apoptosis or necrosis in treated as compared to untreated tumors and on expression of p21, p27, EGFR and phospho-EGFR in aerodigestive tract tumors.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have pathological confirmation of non small cell carcinoma of the aerodigestive tract (lung, esophagus, head and neck cancer).
* Patients must have resectable clinical stage I - III non small cell lung, clinical stage I-III esophageal cancer, or stage I-IV A head and neck cancer.
* Age >18 years.
* Adequate hepatic and renal function documented prior to study entry to include: hepatic transaminases (AST or ALT) ≤ 2.0 times the upper limits of normal, total bilirubin ≤ 1.5 times the upper limits of normal, serum creatinine ≤ 1.5 times the upper limit of normal or estimated creatinine clearance ≥ 60 mL/min.
* All patients must be medical candidates for surgical resection of their non-small cell lung cancer.
* All patients must give informed consent indicating they are aware of the investigational nature of this treatment.

Exclusion Criteria:

* Patients may not have received radiation therapy for their aerodigestive tract cancer.
* Patients may not have received chemotherapy for their aerodigestive tract cancer.
* Women must be surgically sterilized or post-menopausal or women of childbearing potential must be using an adequate method of contraception. Women of childbearing potential must be using at least one of the following: oral, implanted, injectable contraceptive hormones, or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or have a partner that is sterile (e.g., vasectomy). Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to start of study therapy.
* Women who are pregnant or breast-feeding will be excluded.
* Male patients with partners of childbearing potential not using an adequate method of birth control as described in the previous paragraph will be excluded.
* Patients with gastrointestinal abnormalities including: inability to take oral medication, requirement for intravenous alimentation, or prior surgical procedures affecting absorption will be excluded.
* A serious uncontrolled medical disorder or active infection which would impair their ability to receive study treatment will be excluded. Significant cardiac disease, including uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous 3 months or serious cardiac arrythmias will be excluded. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol will be excluded.
* Patients with active HIV, Hepatitis C virus (HCV) or Hepatitis B virus (HBV) infection.
* No prior treatment with histone deacetylase (HDAC) inhibitors. Valproic acid is acceptable if not used as anticancer therapy and a 30-day wash-out period is allowed.
* Exposure to other investigational agents within 30 days of study inclusion
* Patients with a "currently active" second malignancy, other than nonmelanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled. Patients would not be considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >5 years or are considered by their physician to be at less than 30% risk of relapse.
* Patients with history of pulmonary embolism who are not receiving anticoagulation, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin H. Dragnev, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with clinical Stage I, II, III A NSCLC or Stage I, II , III esophageal cancer or Stage I, II, III, IV A Head and Neck cancer and a pre-treatment biopsy having at least 3 unstained slides were eligible. Patients were recruited from the oncology clinic.
Groups:
- Vorinostat: Vorinostat 400mg one daily administered orally for 7 to 10 days prior to a second biopsy/ thoracotomy.
Period: Overall Study
Arm/Group | Vorinostat
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat: Vorinostat group
Arm/Group | Vorinostat
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (17.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in Tumor Markers on Tumors of the Lung, Esophagus, or Head and Neck, After 7 Days of Treatment With Vorinostat
Description: Immunohistochemical score, defined as: 0, no tumor cells staining positive; 1+, 0% to 50% of tumor cells staining positive; 2+, 50% to 75% of tumor cells staining positive; and 3+, 75% to 100% of tumor cells staining positive. The change in the score before and after treatment is percentage - 0-100
Time Frame: Baseline to Day 7
Population: Participants who had at least two days days of treatment with vorinostat.
Measure: Median (95% Confidence Interval); unit: percentage of change
Groups:
- Vorinostat: Vorinostat 400 mg once daily orally for 7 to 10 days prior to a second biopsy/ thoracotomy.
Arm/Group | Vorinostat
Number analyzed (Participants) | 10
percentage of change
  Changes in Ki-67 expression by immunohistochemical | 67 [0 to 88]
  Changes in cyclin D1 expression by immunohistochem | 40 [0 to 87]
  Changes in cyclin E expression by immunohistochemi | 40 [0 to 50]

2. Secondary Outcome: Concentration of Vorinostat in Tumor Tissue
Description: Concentration of vorinostat in tumor tissue will be measured after 7 days of use of Vorinostat.
Time Frame: Day 7 from Baseline
Measure: Median (95% Confidence Interval); unit: ng/mg
Groups:
- Vorinostat Intratumoral Concentrations: Vorinostat 400mg one daily administered orally for 7 days prior to a second biopsy/ thoracotomy.
Arm/Group | Vorinostat Intratumoral Concentrations
Number analyzed (Participants) | 10
ng/mg | 42.6 [0 to 80.3]

3. Secondary Outcome: Effects of Vorinostat Treatment on Induction of Apoptosis or Necrosis in Treated vs. Untreated Tumors
Description: vorinostat's effects on induction of apoptosis or necrosis in treated vs untreated tumors and on p21, p27, EGFR, and phospho-EGFR expression aerodigestive tract tumors. Immunohistochemical score is defined as follows: 0, no tumor cells staining positive; 1+, 0% to 50% of tumor cells staining positive; 2+, 50% to 75% of tumor cells staining positive; and 3+, 75% to 100% of tumor cells staining positive.
Time Frame: Baseline to day 7
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Necrosis: Vorinostat 400mg one daily administered orally for 7 days prior to a second biopsy/ thoracotomy.
Arm/Group | Necrosis
Number analyzed (Participants) | 10
score on a scale | 1 [0 to 3]

ADVERSE EVENTS:
Arm/Group | Vorinostat
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Patients were asked to take vorinostat for at least 7 days with a maximum of 10 days. Two participants did not follow directions correctly and took the pills for 3 days and 2 days. One participant took medication at 100mg per day and not the 400 mg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No